CLINICAL TRIAL: NCT03841682
Title: Engaging Self-Regulation Targets to Understand the Mechanism of Behavior Change and Improve Mood and Weight Outcomes- Second Phase (ENGAGE-2)
Brief Title: Engaging Self-regulation Targets to Improve Mood and Weight and Understand Mechanism in Depressed and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Stanford University (Other); University of Washington (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jun Ma, Professor of Medicine, Director of Center for Health Behavior Research, MD, PhD, FAHA, FABMR, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-1174; UH3HL132368 (NIH)
Record Dates: First submitted 2019-02-02; First posted 2019-02-15 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Obesity; Depression
MeSH Terms: conditions — Obesity; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-CARE2 Intervention (Experimental): Participants should continue with their usual medical care. Additionally, participant receive the I-CARE2 intervention.
  Trained health coaches deliver the I-CARE2 intervention over 6 months. The intervention provides 9 individual counseling sessions on problem solving treatment and behavior counselling to manage mood and lose weight (4 weekly, 2 biweekly, and then 3 monthly; 1 hour each), 11 home-viewed GLB videos (weekly; 20-30 minutes each), and self-study and self-monitoring activities. Throughout the intervention, participants are asked to wear and sync a study-provided Fitbit pedometer, and to log their weight, minutes of physical activity, and dietary intake using the Fitbit website or mobile app.
  Interventions: Behavioral: I-CARE2
- Usual Care (No Intervention): Participants should continue with their Usual Medical Care. Additionally, participants receive information on wellness and behavioral health promotion at UI Health and a Fitbit pedometer.

INTERVENTIONS:
Behavioral: I-CARE2 — I-CARE2 intervention synergistically integrates 2 proven national programs: the Program to Encourage Active and Rewarding Lives (PEARLS) for depression care and the Group Lifestyle Balance (GLB) program for weight loss and cardiometabolic risk reduction.
  The PEARLS program provides problem-solving therapy (PST) as first-line for treating depression, with as-needed antidepressant medication intensification. Adapted from the original Diabetes Prevention Program, the GLB program promotes healthy lifestyle change for weight loss and increased physical activity.
  Arms: I-CARE2 Intervention

SUMMARY:
Multimorbidity (i.e., the coexistence of 2 or more chronic conditions in an individual) is increasingly recognized as a pressing public health problem. Effective interventions targeting coexisting depression and obesity are critical given the high prevalence and worsened outcomes for patients with both conditions.

ENGAGE-2 is a pilot randomized controlled trial (RCT). The objective is to investigate the outcomes and mechanisms of an integrated depression and obesity intervention that combines collaborative stepped depression treatment and evidence-based behavioral weight loss treatment. The Integrated Coaching for Better Mood and Weight-2 (I-CARE2) intervention synergistically integrates 2 proven national programs: the Program to Encourage Active and Rewarding Lives (PEARLS) for depression care and the Group Lifestyle Balance (GLB) program for weight loss and cardiometabolic risk reduction.

In Phase 1 of the ENGAGE project, investigators developed a new protocol to quantify activation and connectivity of the Affective, Cognitive Control, and Default Mode brain circuits from functional magnetic resonance imaging (fMRI) among 108 depressed obese patients. Investigators implement the same fMRI protocol in this second phase of the project to examine the mechanistic role of these brain circuits as potential neural targets in treatment engagement and response in the I-CARE2 intervention. A new sample of 105 depressed obese patients are randomized in a 2:1 ratio to receive the I-CARE2 intervention (n=70) or usual care (n=35). Study assessments occur at 0 (baseline), 2 and 6 months. Investigators hypothesize that 1 or more of the neural targets under study will moderate (baseline state) and/or mediate (change at follow-up) the effect of the I-CARE2 intervention versus usual care on health behaviors (problem-solving ability, dietary intakes, physical activity) and clinical outcomes (weight loss, depression, anxiety).

DETAILED DESCRIPTION:
Participants in this study are adult patients with comorbid depression and obesity from outpatient clinics in the University of Illinois Hospital and Health Sciences System (UI Health). Participants will be randomly assigned to receive intervention or usual care control.

The I-CARE2 intervention synergistically integrates the PEARLS program for depression care the GLB program for weight loss. The PEARLS program provides problem-solving therapy (PST) as first-line for treating depression, with as-needed antidepressant medication intensification. Adapted from the original Diabetes Prevention Program, the GLB program promotes healthy lifestyle change for weight loss and increased physical activity. For combination treatment, the I-CARE2 intervention provides 9 individual counseling sessions (4 weekly, 2 biweekly, and then 3 monthly; 1 hour each) and participant self-study materials (GLB videos, handouts, weight and activity tracking) over 6 months.

In response to the funding mechanism for this project, the specific aim of the ENGAGE-2 pilot study is to test the degree to which engaging the validated self-regulation target(s) produces desired behavior change important for weight management and mood.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years
* Body mass index based on study measurements at baseline group orientation: ≥30.0 kg/m2 (≥27.0 if Asian), and weight <350 pounds (due to fMRI scanner size limitations)
* Elevated depressive symptoms as per 9-item Patient Health Questionnaire (PHQ-9) scores ≥10 on study screening
* UI Health patient seen in primary care at least once in the preceding 18 months
* Able and willing to enroll and provide written informed consent

Exclusion Criteria:

* Active suicidal ideation based on PHQ-9 or the 20-item depression symptom checklist (SCL-20) that includes active plan and/or intent
* Any other psychiatric disorder other than persistent depressive disorder and/or major depressive disorder, with the exception of any comorbid anxiety disorder
* Active Bulimia Nervosa within the past 3 months (however Binge Eating Disorder without purging is not an exclusionary condition)
* Active alcohol or substance use disorder (including prescription drugs)
* Currently under the care of a psychiatrist or licensed mental health therapist outside of UI Health
* Had bariatric surgery (e.g., bypass, banding, sleeve, or biliopancreatic diversion with duodenal switch) within the past 12 months or plan to undergo bariatric surgery during the study period
* Pre-existing diabetes (other than during pregnancy)
* Pre-existing cardiovascular disease: e.g., coronary heart disease (myocardial infarction, angina pectoris, percutaneous coronary intervention, and coronary artery bypass graft surgery), cerebrovascular disease (stroke, transient ischemic attack), peripheral vascular disease, heart failure, or aortic aneurysm.
* Diagnosis of cancer (other than non-melanoma skin cancer) that is/was active or treated with radiation or chemotherapy within the past year
* Severe medical comorbidities that require aggressive treatment, e.g., stage 4 or greater renal disease, and liver failure
* Diagnosis of a terminal illness and/or residence in a long-term care facility
* Cognitive impairment based on the Callahan 6-item screener
* MRI is contraindicated (weight over 350 pounds, traumatic brain injury, tumor or any other known structural abnormality in brain, bullet, shrapnel, or other projectile above the shoulder, not being able to lie down in an fMRI scanner for about an hour due to claustrophobia, personal history of epilepsy, convulsions, or seizures, have piercings that cannot be removed)
* Traumatic brain injury; Tumor or any other known structural abnormality in brain
* Inability to speak, read or understand English
* No reliable telephone service, or no regular Internet access via a computer and/or mobile device (e.g., smartphone)
* Plan to move out of the area or transfer care outside UI Health during the study period
* Currently pregnant, lactating, or planning to become pregnant during the study period
* Already enrolled, or planning to enroll, in another medical or behavioral intervention research study
* Family/household member of another participant or of a staff member
* Investigator discretion for clinical safety or protocol adherence reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Depression Symptom Checklist 20 items (SCL-20) at 6 months | Baseline, 6 months
  The SCL-20 is a valid, reliable measure of depression severity, scores ranging from 0 (best) to 4 (worst). SCL-20 cutoff points of 1.5 and 2.0 correspond to moderate and severe depression, respectively. It has been used in numerous depression treatment trials in primary care and community settings, making it particularly useful for cross-study comparisons and data synthesis in meta-analyses.
Change in Boby Mass Index (BMI) at 6 months | Baseline, 6 months
  BMI will be calculated based on height and weight measured per standard protocols

SECONDARY OUTCOMES:
Anxiety | Baseline, 6 months
  Anxiety is measured using Panic Disorder module of the Mini-International Neuropsychiatric Interview (MINI).
Self-regulation of emotion, cognition, and self-reflection | Baseline, 2 months, 6 months
  fMRI scan will be used to evaluate self-regulation of emotion, cognition, and self-reflection
Change in Depression Symptom Checklist 20 items (SCL-20) at 2 months | Baseline, 2 months
  The SCL-20 is a valid, reliable measure of depression severity, scores ranging from 0 (best) to 4 (worst). SCL-20 cutoff points of 1.5 and 2.0 correspond to moderate and severe depression, respectively. It has been used in numerous depression treatment trials in primary care and community settings, making it particularly useful for cross-study comparisons and data synthesis in meta-analyses.
Change in Body Mass Index (BMI) at 2 months | Baseline, 2 months
  BMI will be calculated based on height and weight measured per standard protocols
Anxiety | Baseline, 2 months, 6 months
  Anxiety is measured using Generalized Anxiety Disorder Scale (GAD-7).
Dietary Intake | Baseline, 2 months, 6 months
  Dietary intake will be recorded using 24-hours dietary recalls
Fruit, vegetable, fat and fiber intake | Baseline, 2 months, 6 months
  17-item fruit, vegetable, fat, and fiber screener will be used.
Physical activity (PA) | Baseline, 2 months, 6 months
  PA will be measured using 7-day Physical Activity Recall
Steps | Baseline, 2 months, 6 months
  Steps will be calculated using Fitbit
Problem solving | Baseline, 2 months, 6 months
  Problem Solving will be evaluated using Social Problem-Solving Inventory-Revised: Short Form
Depression Response | 2 months, 6 months
  This will be evaluated using depression symptom checklist SCL-20 (50% decline in SCL-20 scores from baseline)
Complete Depression Remission | 2 months, 6 months
  Evaluated using depression symptom checklist SCL-20 (SCL-20 <0.5)
Weight (kg) | Baseline, 2 months, 6 months
  Measured using a weight scale. Missing study-measured weight may be replaced with weight from electronic health records or self-reported weight.
Clinically significant weight change from baseline | 2 months, 6 months
  Dichotomous variable based on if participants reaching 5% weight loss from baseline.
Blood pressure | Baseline, 2 months, 6 months
  The American Heart Association recommendations for BP measurement will be followed. BP will be measured in the seated position after at least a 5-minute rest in a separate, quiet room where no other activity is taking place and where temperature fluctuations are minimal. At baseline, both arms will be measured once and 2 more times on the arm with higher systolic reading using standard equipment. This same arm will be measured 3 times at each follow-up assessment. Wait 1 minute between each measurement.
Waist circumference | Baseline, 2 months, 6 months
  Waist circumference will be measured using a study-provided body tape measure placed on bare skin in a horizontal plane around the abdomen at the uppermost lateral border of the right iliac crest. Waist circumference will be measured to the nearest 0.1 centimeters. Two measurements will be taken, and if the measurements differ by 1.0 cm or more, then take a third.
Sleep and wake function | Baseline, 2 months, 6 months
  Sleep quality will be assessed on the 8-item Patient-Reported Outcomes Measurement Information System (PROMIS™) sleep disturbance (SD) and sleep-related impairment (SRI) scales short forms. The former measures symptoms of insomnia and the latter measures symptoms of daytime sleepiness. Each item is scaled from 1 (not at all) to 5 (very much). Correlation between the SD short form and the Pittsburgh Sleep Quality Index (PSQI, hypothesized to measure similar attributes) is 0.83 and correlation between the SRI short form and the Epworth Sleepiness Scale (ESS, hypothesized to measure a related but slightly different construct, the propensity to doze during activities) is 0.46, similar to the correlations between the SD full banks and PSQI (0.85) and between SRI full banks and the ESS (0.45).
Perceived stress | Baseline, 6 months
  Perceived stress is measured using Perceived stress scale (PSS). PSS measures the perception of stress (i.e., the degree to which situations in one's life are appraised as stressful). PSS contains 14 items, rated on a 5-point scale ranging from "never" to "very often." After reversing the scores on 7 positive items, a sum of score is calculated with higher score indicating higher perceived stress. Cronbach's alpha ranged from 0.84 to 0.86.
Disability | Baseline, 6 months
  Disability is measured using Sheehan Disability Scale. The Sheehan Disability Scale is a validated questionnaire that measures functional disability and is sensitive to treatment effects in clinical trials. Patients rate the extent to which their symptoms impair work/school, social, and family life on a visual analog scale from0 to 10 and answer the number of days when their symptoms cause them to miss work/school and be unproductive at work/school.
Generic health related quality of life | Baseline, 6 months
  Generic health related quality of life is measured using SF-8 Health Survey. The SF-8 is an 8-item version of the SF-36 that measures overall health-related quality of life. Physical and mental health composite scores are computed using the scores of 8 questions and range from 0 to 100, with 0 indicating the lowest level of health and 100 indicating the highest level of health. Correlation between the SF-8 and the SF-36 is 0.825 for physical health component and 0.881 for mental health component.
Obesity-specific health related questions | Baseline, 6 months
  The Obesity-Related Problem Scale specifically measures the impact of obesity on psychosocial functioning. The 8-item scale has high internal reliability and sound test-retest reliability, correlates strongly with a wide range of theoretically related constructs, and is responsive to weight loss intervention.
Posttraumatic stress disorder | Baseline, 6 months
  Posttraumatic stress disorder is measured using the 17-item PTSD checklist - Civilian Version (PCL-C) that has high reliability and validity.
Pain interference and intensity | Baseline, 6 months
  Pain is measured using PROMIS SF - Pain Interference 4a and Numeric Rating Scale - Pain Intensity 1a.
Binge eating severity | Baseline, 6 months
  Binge eating severity is measured using the Binge eating severity scale.
Use of general wellness programs and services questionnaire | 6 months
  This questionnaire asks participants if they have received a list of wellness programs and services for general physical and mental well-being in the past 6 months.
Self-regulation of emotion, cognition, & self-reflection | Baseline, 2 months, 6 months
  BiAffect (Smart phone passive data collection) will be used, as an alternative, to evaluate self-regulation of emotion, cognition, and self-reflection

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, MD,PhD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - Institute for Health Research and Policy (IHRP), Center for Health Behavior Research, Chicago, Illinois
  - UIMC Advanced Imaging Center, Chicago, Illinois

REFERENCES:
- [Derived] Lv N, Hallihan H, Xiao L, Williams LM, Ajilore OA, Ma J. Association of Changes in Neural Targets and Dietary Outcomes among Patients with Comorbid Obesity and Depression: Post hoc Analysis of ENGAGE-2 Mechanistic Clinical Trial. J Nutr. 2023 Mar;153(3):880-896. doi: 10.1016/j.tjnut.2023.01.022. Epub 2023 Jan 23. PMID 36931755
- [Derived] Burton TC, Lv N, Tsai P, Penalver Bernabe B, Tussing-Humphreys L, Xiao L, Pandey GN, Wu Y, Ajilore OA, Ma J. Associations between fecal short-chain fatty acids, plasma inflammatory cytokines, and dietary markers with depression and anxiety: Post hoc analysis of the ENGAGE-2 pilot trial. Am J Clin Nutr. 2023 Apr;117(4):717-730. doi: 10.1016/j.ajcnut.2023.01.018. Epub 2023 Feb 1. PMID 36796440
- [Derived] Kannampallil T, Dai R, Lv N, Xiao L, Lu C, Ajilore OA, Snowden MB, Venditti EM, Williams LM, Kringle EA, Ma J. Cross-trial prediction of depression remission using problem-solving therapy: A machine learning approach. J Affect Disord. 2022 Jul 1;308:89-97. doi: 10.1016/j.jad.2022.04.015. Epub 2022 Apr 7. PMID 35398399
- [Derived] Lv N, Ajilore OA, Ronneberg CR, Venditti EM, Snowden MB, Lavori PW, Xiao L, Goldstein-Piekarski AN, Wielgosz J, Wittels NE, Barve A, Patel AS, Eckley TL, Stetz P, Gerber BS, Smyth JM, Simmons JM, Rosas LG, Williams LM, Ma J. The ENGAGE-2 study: Engaging self-regulation targets to understand the mechanisms of behavior change and improve mood and weight outcomes in a randomized controlled trial (Phase 2). Contemp Clin Trials. 2020 Aug;95:106072. doi: 10.1016/j.cct.2020.106072. Epub 2020 Jul 2. PMID 32621905